CLINICAL TRIAL: NCT01203384
Title: Placebo-Controlled, Ascending Multiple-Dose Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of CHF5074 in Healthy Young Male Subjects
Brief Title: Study to Evaluate Safety, Pharmacokinetics and Pharmacodynamics of CHF5074 in Healthy Young Male Subjects
Acronym: CT02
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CERESPIR (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCD-0913-PR-0038
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- CHF5074 1x (Experimental): oral tablet, multidose
  Interventions: Drug: CHF5074 1x
- CHF5074 2x (Experimental): oral tablet, multidose
  Interventions: Drug: CHF5074 2x
- CHF5074 3x (Experimental): oral tablet, multidose
  Interventions: Drug: CHF5074 3x
- Placebo (Placebo Comparator): placebo, oral tablet, multidose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CHF5074 1x — oral tablet, 1x, once a day in the morning for 14 days
  Arms: CHF5074 1x
Drug: CHF5074 2x — oral tablet, 2x, once a day in the morning for 14 days
  Arms: CHF5074 2x
Drug: CHF5074 3x — oral tablet, 3x, once a day in the morning for 14 days
  Arms: CHF5074 3x
Drug: Placebo — oral tablet, placebo, once a day in the morning for 14 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of multiple oral doses of CHF5074 in young healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Subject is judged to be in good health on the basis of medical history, complete physical examination including vital signs, 12-lead electrocardiogram (ECG) and standard laboratory tests.

Exclusion Criteria:

* Medical history (within the last 10 years) of major cardiovascular, hepatic or renal disease.
* Abnormal results of liver function tests, renal function tests or thyroid tests performed at screening.
* Significant allergic conditions that require medical treatment
* Use of any psychoactive, recreational or prescription drug within the 4 weeks prior to study drug administration.
* Use of ibuprofen, sulindac sulfide, indomethacin, flurbiprofen within 2 weeks prior to study drug administration.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2010-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Adverse Events | from Screening through Day 18

SECONDARY OUTCOMES:
Dose linearity of CHF5074 plasma levels (Cmax) | Day -1 through Day 18
Dose linearity of CHF5074 plasma levels (AUC 0-t) | Day -1 through Day 18

CONTACTS AND LOCATIONS:
Overall Officials: Magdy L Shenouda, MD, Principal Investigator — Iberica Clinical Research Center
Locations (1):
- Iberica Clinical Research Center, Eatontown, New Jersey, United States